CLINICAL TRIAL: NCT02847715
Title: Electronic Patient Self-Reported Outcomes to Improve Cancer Management and Patient Experiences: Implement the System for Remote Monitoring of Cancer Patients in Remission
Brief Title: Electronic Patient Self-Reported Outcomes to Improve Cancer Management and Patient Experiences
Acronym: ePRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Yorkshire Cancer Research (Other); The Leeds Teaching Hospitals NHS Trust (Other); Bradford Teaching Hospitals NHS Foundation Trust (Other Government); Calderdale and Huddersfield NHS Foundation Trust (Other); Airedale NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Galina Velikova, Professor of Psycho-social and Medical Oncology/Consultant in Medical Oncology, University of Leeds
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: L392 (gynae)
Record Dates: First submitted 2016-05-19; First posted 2016-07-28 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cancer
Keywords: PRO; PROM; Adverse event; QTool; Aftercare
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Audit phase (No Intervention): In the audit-phase, a group of 59 patients will be recruited and followed over a 12 month period. Data will be collected on clinical and patient outcomes in an audit in order to be able to compare to the intervention (after-phase) group.
- Intervention (pilot-phase) (Experimental): In the pilot-phase, a group of 59 patients will be recruited and followed over a 6-12 month period. Patients in this group will be assigned to the new remote monitoring follow-up pathway (ePRIME), whereby instead of attending routine outpatient appointments they are monitored remoted via a online symptom monitoring questionnaire and related clinical tests undertaken remotely. All information is collated in the patient's electronic patient record, and clinicians will review/respond to the data as necessary.
  Interventions: Device: ePRIME

INTERVENTIONS:
Device: ePRIME — ePRIME is an remote monitoring pathway that includes an online system for patients to self-report symptoms and AE following cancer treatments. ePRIME allows AE reporting from home and enables patient reported data to be integrated into existing EPR to allow for the reports to be used in routine care. In addition the system is capable of generating alerts for serious symptoms to the relevant clinical team and providing patient advice on managing mild and moderate symptoms.
  Arms: Intervention (pilot-phase)

SUMMARY:
Improvements in cancer treatment have led to an increasing number of patients being cured or in remission, but they are followed up to detect recurrence, manage persistent symptoms and late treatment effects. With growing survivors, traditional hospital follow-up is not sustainable. New models of follow-up care are needed. This research project aims to develop and establish the feasibility of introducing a new electronic care pathway/system for remote monitoring ovarian cancer patients in remission. The project includes a development phase, followed by an audit & pilot intervention phase to explore the feasibility of a new pathway/system for remote monitoring.

DETAILED DESCRIPTION:
Background Improvements in cancer treatment have led to an increasing number of patients being cured or in remission, but they are followed up to detect recurrence, manage persistent symptoms and late treatment effects. With growing survivors, traditional hospital follow-up is not sustainable. New models of follow-up care are needed.

Aim To develop and establish the feasibility of introducing a new electronic care pathway/system for remote monitoring ovarian cancer patients in remission.

Methods An existing online patient symptom reporting system will be extended for use in remote follow-up. A tracking program will be developed and IT systems integrated in the local hospitals.

Development Phase:

a) Scoping literature review of existing validated symptom measures. b) Consultation with expert groups to establish choice of questions, relevant symptoms, timing/frequency for monitoring. c) Interviews with patients and clinicians to explore current pathway and redesign.

Audit of usual care phase In this phase consecutive eligible ovarian, fallopian tube, primary peritoneal, endometrial or female genital (not otherwise specified) cancer patients (on completion of their first/second line of treatment) will be approached and data on clinical outcomes collected at the routine 3 monthly outpatient appointments for 12 months and PROMs collected 6 monthly. We aim to recruit around 60 patients.

Pilot Intervention phase In the intervention group the feasibility of the re-designed care pathway (intervention) will be piloted in a separate group of eligible ovarian, fallopian tube, primary peritoneal, endometrial or female genital (not otherwise specified) cancer patients. The patients approached will be a mixture of those who are entering follow-up after recently completing their first/second line treatment, and those who have already been attending for some time (months/years) for routine follow-up after their first/second line treatment. We aim to recruit around 60 patients. Consenting patients will be reminded to use the online system every 3 months and have a mandatory blood test by their GP/local hospital. Information will be available for the clinical teams to access electronically. Patients will always have the option to choose to speak or see their 'key clinician'. Virtual clinics will be held for key clinicians to review and respond to remote monitoring data. Clinical and patient outcomes will be collected for a 6-12 month period (this timeframe is dependent on the date of study entry and the funding period remaining). Following the pilot intervention period, 10 patients (or more if deemed necessary) and 6 clinicians will also be interviewed.

Outcomes

* Develop a new electronic care pathway/system for remote monitoring patients in remission
* Obtain initial data on clinical and patient feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or over) attending St James' University Hospital Bexley Wing, Bradford Teaching Hospitals NHS Foundation Trust, Calderdale & Huddersfield NHS Foundation Trust, and Airedale NHS Foundation Trust with stage 2-4 ovarian/fallopian/peritoneal/endometrial cancer in remission following the end of first or second line chemotherapy or end of maintenance Avastin/Bevacizumab (where indicated)
* Patients may have recently completed treatment or already been on routine clinic-based face-to-face follow-up at the time of recruitment into the pilot intervention phase
* Able and willing to give informed consent
* Able to read and understand English
* Access to the internet

Exclusion Criteria:

* Exhibiting overt psychopathology/cognitive dysfunction
* Taking part in other clinical trials involving the completion of extensive patient reported outcome or quality of life measures or requiring scheduled face-to-face clinical outpatient appointments (Intervention group only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients recruited / Number of patients approached (=consent rate) | Baseline
  Number of patients recruited and number of patients approached will be logged by research team during recruitment (including reasons for non-recruitment)
Number of participant withdrawals | 12 months
  Number of participant withdrawals will be logged by research team at the time of any withdrawals
Reasons for participant withdrawals | 12 months
  Reasons for withdrawal will be assessed via case record form completed by researcher with the participant at time of withdrawal and collated at the end of the study
Number of participants with self-reported symptom data (questionnaire) at 3 months | 3 months
  Patients will be reminded to complete an electronic questionnaire about their symptoms at 3 months
Number of participants with self-reported symptom data (questionnaire) at 6 months | 6 months
  Patients will be reminded to complete an electronic questionnaire about their symptoms at 6 months
Number of participants with self-reported symptom data (questionnaire) at 9 months | 9 months
  Patients will be reminded to complete an electronic questionnaire about their symptoms at 9 months
Number of participants with self-reported symptom data (questionnaire) at 12 months | 12 months
  Patients will be reminded to complete an electronic questionnaire about their symptoms at 12 months
Patient acceptability (questionnaire/interviews) | 12 months
  Patient acceptability explored through end-of-study questionnaires and interviews
Clinician acceptability (questionnaire/interviews) | 12 months
  Clinician acceptability explored through end-of-study questionnaires and interviews

CONTACTS AND LOCATIONS:
Overall Officials: Galina Velikova, Principal Investigator — University of Leeds
Locations (1):
- St James University Hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kennedy F, Shearsmith L, Holmes M, Velikova G. 'It made me feel part of the team, having my homework to do' - women and specialist nurse experiences of remote follow-up after ovarian cancer treatment: a qualitative interview study. Support Care Cancer. 2022 Dec 13;31(1):2. doi: 10.1007/s00520-022-07470-z. PMID 36512093
- [Derived] Kennedy F, Shearsmith L, Holmes M, Rogers Z, Carter R, Hofmann U, Velikova G. Electronic patient-reported monitoring of symptoms during follow-up of ovarian cancer patients: a feasibility study. BMC Cancer. 2022 Jul 2;22(1):726. doi: 10.1186/s12885-022-09817-5. PMID 35780095
- See also: Research group website/webpage relating to the study — http://www.pogweb.org/index.php/eprime/